CLINICAL TRIAL: NCT05242042
Title: A Multicenter, Double-blind, Randomized, Placebo-Controlled, Phase II/III Study to Evaluate the Efficacy, Safety and Pharmacokinetics of JT001 (VV116) for the Early Treatment of Coronavirus Disease 2019 (COVID-19) in Participants With Mild to Moderate COVID-19.
Brief Title: JT001 (VV116) for the Early Treatment of COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Based on the current number of COVID-19 cases and the approval of COVID-19 treatment drugs , the research team is facing great challenges, and it is decided to terminate this study
Sponsor: Shanghai JunTop Biosciences Co., LTD (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JT001-004-II/III-COVID-19
Record Dates: First submitted 2022-02-11; First posted 2022-02-16 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Mild to Moderate COVID-19
MeSH Terms: interventions — GS-621763

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: JT001
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JT001 — JT001 administered orally in tablet form every 12 hours for 5 days (10 doses total)
  Other Names: VV116
  Arms: Arm 1
Drug: Placebo — Placebo matching JT001 administered orally in tablet form every 12 hours for 5 days (10 doses total)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of JT001 (VV116) for the early Treatment of Coronavirus Disease 2019 (COVID-19) in participants with mild to moderate COVID-19, at high risk for progression to severe COVID-19, including death.

DETAILED DESCRIPTION:
Screening Interested participants will sign the appropriate informed consent form (ICF) prior to completion of any study procedures.

The investigator will review symptoms, risk factors and other non-invasive inclusion and exclusion criteria prior to any invasive procedures. If the participant is eligible after this review, then the site will perform the invasive procedures to confirm eligibility.

Treatment and Assessment Period

* Complete baseline procedures and sample collection
* Participants are randomized to an intervention group
* Participants receive study intervention (Q12H X 5 days)
* Complete all safety monitoring
* Complete all efficacy data collection
* Blood samples collection

ELIGIBILITY:
Inclusion Criteria:

1. Participants of 18 years of age or older
2. Participants who have a positive SARS-CoV-2 test result, and have sample collection for first positive SARS-CoV-2 viral infection determination ≤5 days prior to randomization
3. Participants who have one or more mild or moderate COVID-19 symptoms as follows and have a COVID-19 Related Symptom score ≥3
4. Participants with the onset of symptoms of COVID-19 ≤5 days prior to randomization
5. Participants who satisfy one or more than one of the following high risks for progression to severe COVID-19, including death:
6. Participants who must agree to adhere to contraception restrictions
7. Participants who understand and agree to comply with planned study procedures
8. Participants can give written informed consent approved by the Ethical Review Board governing the site and comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Participants who are judged by the investigator as likely to progress to severe/critical COVID-19 prior to randomization.
2. Participants who have SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300, or respiratory rate ≥30 per minute, or heart rate ≥125 per minute
3. Participants who require mechanical ventilation or anticipated impending need for mechanical ventilation
4. Participants who are suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
5. Participants who have eye disease
6. Participants who have ALT or AST>2 ULN at screening

7 Participants who have known allergies to any of the components used in the formulation of the interventions

8 Any medical condition, which in the opinion of the Investigator, will compromise the safety of the participant

9. Participants who have received a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment) within 180 days prior to screening visit

10. Participants who have received convalescent COVID-19 plasma treatment

11. Participants who have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed

12.Participants who are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

13. Female who is pregnant or breast-feeding or plan to be pregnant within this study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
progression of COVID-19:defined as progress to severe/critical COVID-19 or death from any cause | Up to 28 days
  1. Percentage of the participants who have progression of COVID-19
  2. Time to sustained clinical symptom resolution

SECONDARY OUTCOMES:
Overall participant clinical status | Up to 28 days
  Percentage of participants who experience these events by Day 28
  * Progress to severe COVID-19
  * Progress to critical COVID-19
  * Death from any cause
COVID-19-related hospitalization rate of non-hospitalized participants | Up to 28 days
  Percentage of participants who experience COVID-19-related hospitalization by Day 28
SARS-CoV-2 negative rate through Day7 | Baseline through Day 7
  Percentage of participants who achieve SARS-CoV-2 negative at Day 5 and 7
The plasma concentration | Baseline through Day 5
  The plasma concentration of JT001 (VV116) and major metabolites
Safety assessments | Up to 28 days
  Safety assessments such as AEs and SAEs
SARS-CoV-2 viral load | Baseline through Day 7
  The SARS-CoV-2 viral load change from baseline to Day 5 and 7
SARS-CoV-2 viral load | Baseline through Day 7
  SARS-CoV-2 viral load area under the response time curve (AUC) assessed through Day 7
To assess SARS-CoV-2 viral genetic variation | Day 1
  SARS-CoV-2 viral genetic variation

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ma, Medical Director, Study Director — Shanghai JunTop Biosciences Co., LTD
Locations (8):
- China (6):
  - Chongqing Public Health Medical Center, Chongqing, Chongqing Municipality
  - Thesixth peoples Hospital Of ZhengZhou, Zhengzhou, Henan
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - The Ninth Hospital of Nanchang, Nanchang, Jiangxi
  - The Sixth People's Hospital of ShenYang, Shenyang, Liaoning
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
- Hong Kong (2):
  - CUHK Medical Centre, Hong Kong
  - CUHK Phase 1 Clinical Trial Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Undecided